CLINICAL TRIAL: NCT03903926
Title: Phase Ⅳ Clinical Trial, to Evaluate the Efficacy of the Enterovirus 71 (EV71) Inactivated Vaccine and Its Correlation With EV71 Antibody Level
Brief Title: Efficacy Trial of a Commercial EV71 Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO-EV71-4013
Record Dates: First submitted 2019-03-29; First posted 2019-04-04 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Hand, Foot and Mouth Disease
Keywords: EV71 vaccine; Efficacy; Seroprotective correlates
MeSH Terms: conditions — Hand, Foot and Mouth Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort one (Experimental): 5000 volunteers (6-35 months)-EV71 vaccine
  Interventions: Biological: 5000 volunteers (6-35 months)-EV71 vaccine
- Cohort two (No Intervention): 10000 unvaccinated volunteers (6-35 months)
- Cohort three (No Intervention): 500 unvaccinated volunteers (36-71 months)

INTERVENTIONS:
Biological: 5000 volunteers (6-35 months)-EV71 vaccine — two doses EV71 vaccines will be administrated on day 0, 30 respectively
  Arms: Cohort one

SUMMARY:
The purpose of this post-marketing study is to evaluate the efficacy, immunogenicity, and safety of the EV71 vaccine post marketing, and explore the protective levels of various enterovirus neutralizing antibodies

DETAILED DESCRIPTION:
This study is a post-marketing aims to evaluate the efficacy, immunogenicity, and safety of the EV71 vaccine, and explore the protective levels of various enterovirus neutralizing antibodies. This study includes the following three sections: (1) efficacy study of EV71 vaccine based on enhanced cases monitoring, using prospective cohort study design (2) study on correlation between EV71 vaccine protection and EV71 antibody levels, using case-control study design (3) pathogenic spectrum and sero-epidemiological investigation of hand, foot and mouth disease (HFMD) in children. 15500 volunteers aged 6-71 months are expected to participate in this study, among which 5000 volunteers aged 6-35 months will receive two doses EV71 vaccine manufactured by Sinovac Biotech Co., Ltd, and constitute the experimental cohort. 10000 unvaccinated volunteers aged 6-35 months will constitute the the control cohort. The efficacy evaluation will be conducted based on the abovementioned two cohort. Enhanced HFMD surveillance system will be established to report the HFMD cases in the abovementioned 2 cohorts, as well as another cohort consisting of 500 volunteers aged 36-71 months. The case surveillance period of this study is one year. Laboratory tests will be conducted for case confirmation.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers aged 6-71 months;
* Guardians of the participants voluntarily to vaccinate the participants with EV71 vaccine at their own expense;
* Guardians of the participants should be capable of understanding the written consent form, and such form should be signed prior to enrollment;
* Complying with the requirement of the study protocol;

Exclusion Criteria:

* History of HFMD prior to the study entry;
* Prior vaccination with EV71 vaccine;
* History of allergy to any vaccine, or any ingredient, excipients and Gentamycin Sulfate of the vaccine, or serious adverse reaction(s) to vaccination, such as urticaria, dyspnea, angioneurotic edema, abdominal pain, etc. (only for 6-35 months old subjects of the vaccinated group) ;
* Congenital malformation, developmental disorders, genetic defects, or severe malnutrition (only for 6-35 months old subjects of the vaccinated group);
* Severe/uncontrollable nervous system disease (epilepsy, seizures or convulsions) or mental illness (only for 6-35 months old subjects of the vaccinated group);
* Autoimmune disease or immunodeficiency/immunosuppressive (only for 6-35 months old subjects of the vaccinated group) ;
* History of asthma, angioedema, diabetes or malignancy (only for 6-35 months old subjects of the vaccinated group);
* Acute disease or acute stage of chronic disease within 7 days prior to study entry (only for 6-35 months old subjects of the vaccinated group);
* Axillary temperature > 37.0 Celsius (only for 6-35 months old subjects of the vaccinated group)；
* Any other factor that suggesting the volunteer is unsuitable for this study based on the opinions of investigators.

Ages: 6 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 15500 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
The efficacy of two doses EV71 vaccine in the 6-35 months old subjects | During the case monitoring period of 1 year
  Vaccine Efficacy (VE)=(incidence difference between vaccinated and unvaccinated group/incidence of vaccinated group)*100%
The seroprotective titers of the EV71 neutralizing antibody in the 6-35 months old subjects | Through study completion, an average of 1 year
  Immune correlates of protection

SECONDARY OUTCOMES:
The incidence of adverse events after the EV71 vaccination in the 6-35 months old subjects | Within 6 months after each dose injection
  Safety index
The seroprotective titers of the CA16, CA6, CA10 neutralizing antibody in the 6-35 months old subjects | Through study completion, an average of 1 year
  Immune correlates of protection
The seropositive rate of the EV71, CA16, CA6, CA10 neutralizing antibody in the 6-71 months old subjects | During the study period, 2 months after the study beginning
  Serum epidemiological index
The geometric mean titer (GMT) of the EV71, CA16, CA6, CA10 neutralizing antibody in the 6-71 months old subjects | During the study period, 2 months after the study beginning
  Serum epidemiological index
The seroconversion rate of the EV71 neutralizing antibody after vaccination in the 6-35 months old subjects | 30 days after two doses
  Immunogenicity index
The geometric mean increase (GMI) of the EV71 neutralizing antibody after vaccination in the 6-35 months old subjects | 30 days after two doses
  Immunogenicity index
Proportions of various pathogens in the confirmed HFMD cases | Through study completion, an average of 1 year
  Pathogen spectrum index

CONTACTS AND LOCATIONS:
Overall Officials: Xuhua Guan, Doctor, Principal Investigator — Hubei Provincial Center for Disease Control and Prevention
Locations (2):
- China (2):
  - Songzi Center for Disease Control and Prevention, Jingzhou, Hubei
  - Xiantao Center for Disease Control and Prevention, Xiantao, Hubei